CLINICAL TRIAL: NCT05045807
Title: Randomised Controlled Trial to Investigate N-nitrosamine Formation After Meat Intake - Pilot Study of the Nitrate INFORMER Studies; Nitrate INFORMER Studies: Is Nitrosamine FORMation dEpenent on souRce
Brief Title: Nitrate INFORMER Nitrosamine Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edith Cowan University (Other)
Collaborators: The University of Western Australia (Other); Flinders University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-02629-BONDONNO(pilot)
Record Dates: First submitted 2021-08-30; First posted 2021-09-16 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Health Risk Behaviors
MeSH Terms: conditions — Health Risk Behaviors | interventions — Meat; Vegetables

STUDY DESIGN:
Intervention Model Description: prospective, mono-centre, randomised, controlled, crossover study
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the interventions, participants, and the investigators responsible for delivering the interventions will be unblinded throughout the trial. However, all researchers performing the laboratory analyses and data analyses will be blinded to the interventions that the participants received until after the data analysis has been performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meat with added nitrate (Experimental): Prosciutto/pancetta/Parma ham/salami (all derived from pork) prepared by a commercial butcher with sodium nitrate as an additive.
  Interventions: Dietary Supplement: Meat with added nitrate
- Meat with added nitrate plus vegetables (Experimental): The same intervention as of Arm "meat with added nitrate" consumed together with mixed vegetables.
  Interventions: Dietary Supplement: Meat with added nitrate plus vegetables

INTERVENTIONS:
Dietary Supplement: Meat with added nitrate — Prosciutto/pancetta/Parma ham/salami (all derived from pork) prepared by a commercial butcher with the sodium nitrate and nitrite as an additive.
  Arms: Meat with added nitrate
Dietary Supplement: Meat with added nitrate plus vegetables — The same intervention as of intervention "meat with added nitrate" consumed together with mixed vegetables.
  Arms: Meat with added nitrate plus vegetables

SUMMARY:
Nitrate is a controversial component of vegetables, meat, and drinking water. The now well-established benefits of nitrate, through the enterosalivary nitrate-nitrite-nitric oxide (NO) pathway, on cardiovascular risk factors and long-term cardiovascular disease risk are tarnished by a continuing concern about a link between nitrate ingestion and cancer. This can result in misguided advice to avoid consumption of high-nitrate leafy green vegetables by both the media and the scientific literature. A recent media headline stated, "Cancer alert over rocket: trendy salad leaves exceed safe levels of carcinogenic nitrates in one in every ten samples". One scientific review stated, "the presence of nitrate in vegetables, as in water and generally in other foods, is a serious threat to man's health". Controversy in the literature, and gaps in the knowledge are leading to confusing messages around vegetables that may play a critical role in cardiovascular health.

The major dietary sources of nitrate are vegetables, meat, and drinking water. Source of nitrate could be a crucial factor determining whether the consumption of nitrate is linked with beneficial (such as improving cardiovascular health) versus harmful (N-nitrosamine formation) effects. For example, unlike meat and water-derived nitrate, vegetables contain high levels of vitamin C and/or polyphenols that may inhibit the production of N-nitrosamines. So far, no study has investigated the formation of N-nitrosamines after consumption of these different sources in humans.

A pilot study will be conducted to determine that endogenous N-nitrosamine formation is observed after ingestion of meat with added nitrate and nitrite and that consumption of vegetables with the meat containing added nitrate and nitrite will inhibit the production of N-nitrosamines.

DETAILED DESCRIPTION:
Study design:

A crossover study design will be used with a 1-week washout period. Each participant will complete the scheduled study visits for one of the dietary interventions which will be assigned in random order. Following the washout, the participants will then complete the scheduled study visits for the remaining intervention. Participants will be provided with a low nitrate and N-nitrosamine meal on the preceding evening of each study visit. These meals will be consistent across all study visits. Participants will be asked to refrain from drinking coffee and any alcoholic beverage and doing any exercise 24 hours prior to the study visit.

Dietary interventions:

Meat with added nitrate: Prosciutto/pancetta/Parma ham/salami (all derived from pork) prepared by a commercial butcher with sodium nitrate as an additive.

Meat with added nitrate plus vegetables: The same intervention described above consumed together with mixed vegetables.

Assessments:

At each clinic visit, baseline samples of urine will be collected for measurement of N-nitrosamines, nitrate, and nitrite. After the intervention, all urine within the first 240 minutes and then subsequent 20-hour period will be collected for measurement of N-nitrosamines, nitrate, and nitrite.

ELIGIBILITY:
Inclusion Criteria:

* Six healthy, ambulant, community-dwelling men and women aged between 18 to 55 years old and with no history of major chronic disease will be recruited from the Perth general population.

Exclusion Criteria:

Individuals volunteering to participate in the study will be excluded according to the following criteria:

* current or recent (<12 months) smoking
* body mass index (BMI) <18 or > 35 kg/m2
* systolic blood pressure > 160 mmHg
* diastolic blood pressure > 100 mmHg
* any major illness such as cancer, psychiatric illness, diagnosed diabetes
* use of any of the following medications: statins, antihypertensives, nitric oxide donors, antithrombotic medication, anti-coagulant medication, anti-arrhythmic drugs, beta-blockers, regular aspirin use, regular proton pump inhibitor use
* alcohol consumption > 30g/day
* who are pregnant, lactating, or wishing to become pregnant during the study
* use of antibiotics within the previous 12 weeks of the study
* regular use of mouthwash and not willing to cease mouthwash use for the duration of the study
* participation on other research studies
* major gastrointestinal tract condition e.g. Crohns disease and inflammatory bowel disease
* and inability or unwillingness to follow the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
N-nitrosamines in urine pre each intervention | At each clinic visit, baseline samples of urine will be collected.
  Participants will be provided with a sterilized container and instructions to collect the first urine sample of the day which will be brought into the clinic. Urine aliquots will be frozen at -80°C until analysis. Level of N-nitrosamines will be measured by gas chromatography mass spectrometry (GCMS).
N-nitrosamines in urine post each intervention up to 240 min | At each clinic visit, all urine samples within the first 240 min will be collected.
  Participants will be provided with a sterilized container and instructions to collect all urine until 4 hours post intervention. Urine aliquots will be frozen at -80°C until analysis. Level of N-nitrosamines will be measured by gas chromatography mass spectrometry (GCMS).
N-nitrosamines in urine post each intervention after 4 hours up till 24 hours | After each clinic visit, all urine from 4-hour to 24-hour period will be collected.
  Participants will be provided with a sterilized container and instructions to collect all urine from 4 hours until 24 hours post intervention. Urine aliquots will be frozen at -80°C until analysis. Level of N-nitrosamines will be measured by gas chromatography mass spectrometry (GCMS).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine P Bondonno, PhD, RNutr., Principal Investigator — Edith Cowan University
Locations (1):
- Royal Perth Hospital Research Foundation, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lundberg JO, Weitzberg E. NO-synthase independent NO generation in mammals. Biochem Biophys Res Commun. 2010 May 21;396(1):39-45. doi: 10.1016/j.bbrc.2010.02.136. PMID 20494108
- [Result] Blekkenhorst LC, Bondonno NP, Liu AH, Ward NC, Prince RL, Lewis JR, Devine A, Croft KD, Hodgson JM, Bondonno CP. Nitrate, the oral microbiome, and cardiovascular health: a systematic literature review of human and animal studies. Am J Clin Nutr. 2018 Apr 1;107(4):504-522. doi: 10.1093/ajcn/nqx046. PMID 29635489
- [Result] Bondonno CP, Blekkenhorst LC, Liu AH, Bondonno NP, Ward NC, Croft KD, Hodgson JM. Vegetable-derived bioactive nitrate and cardiovascular health. Mol Aspects Med. 2018 Jun;61:83-91. doi: 10.1016/j.mam.2017.08.001. Epub 2017 Sep 7. PMID 28802834
- [Result] Spiegelhalder B, Eisenbrand G, Preussmann R. Influence of dietary nitrate on nitrite content of human saliva: possible relevance to in vivo formation of N-nitroso compounds. Food Cosmet Toxicol. 1976 Dec;14(6):545-8. doi: 10.1016/s0015-6264(76)80005-3. No abstract available. PMID 1017769
- [Result] Tannenbaum SR, Weisman M, Fett D. The effect of nitrate intake on nitrite formation in human saliva. Food Cosmet Toxicol. 1976 Dec;14(6):549-52. doi: 10.1016/s0015-6264(76)80006-5. No abstract available. PMID 1017770
- [Result] Gangolli SD, van den Brandt PA, Feron VJ, Janzowsky C, Koeman JH, Speijers GJ, Spiegelhalder B, Walker R, Wisnok JS. Nitrate, nitrite and N-nitroso compounds. Eur J Pharmacol. 1994 Nov 1;292(1):1-38. doi: 10.1016/0926-6917(94)90022-1. PMID 7867685
- [Result] Mirvish SS. Role of N-nitroso compounds (NOC) and N-nitrosation in etiology of gastric, esophageal, nasopharyngeal and bladder cancer and contribution to cancer of known exposures to NOC. Cancer Lett. 1995 Jun 29;93(1):17-48. doi: 10.1016/0304-3835(95)03786-V. PMID 7600541
- [Result] IARC Working Group on the Evaluation of Carcinogenic Risks to Humans. IARC monographs on the evaluation of carcinogenic risks to humans. Ingested nitrate and nitrite, and cyanobacterial peptide toxins. IARC Monogr Eval Carcinog Risks Hum. 2010;94:v-vii, 1-412. No abstract available. PMID 21141240
- [Result] Hord NG, Tang Y, Bryan NS. Food sources of nitrates and nitrites: the physiologic context for potential health benefits. Am J Clin Nutr. 2009 Jul;90(1):1-10. doi: 10.3945/ajcn.2008.27131. Epub 2009 May 13. PMID 19439460
- [Result] Blekkenhorst LC, Prince RL, Ward NC, Croft KD, Lewis JR, Devine A, Shinde S, Woodman RJ, Hodgson JM, Bondonno CP. Development of a reference database for assessing dietary nitrate in vegetables. Mol Nutr Food Res. 2017 Aug;61(8). doi: 10.1002/mnfr.201600982. Epub 2017 May 3. PMID 28105786
- [Result] Bartsch H, Ohshima H, Pignatelli B. Inhibitors of endogenous nitrosation. Mechanisms and implications in human cancer prevention. Mutat Res. 1988 Dec;202(2):307-24. doi: 10.1016/0027-5107(88)90194-7. PMID 3057363
- [Result] Levallois P, Ayotte P, Van Maanen JM, Desrosiers T, Gingras S, Dallinga JW, Vermeer IT, Zee J, Poirier G. Excretion of volatile nitrosamines in a rural population in relation to food and drinking water consumption. Food Chem Toxicol. 2000 Nov;38(11):1013-9. doi: 10.1016/s0278-6915(00)00089-2. PMID 11038239
- [Result] Bartholomew B, Hill MJ. The pharmacology of dietary nitrate and the origin of urinary nitrate. Food Chem Toxicol. 1984 Oct;22(10):789-95. doi: 10.1016/0278-6915(84)90116-9. PMID 6541617
- [Result] Bondonno CP, Croft KD, Puddey IB, Considine MJ, Yang X, Ward NC, Hodgson JM. Nitrate causes a dose-dependent augmentation of nitric oxide status in healthy women. Food Funct. 2012 May;3(5):522-7. doi: 10.1039/c2fo10206d. Epub 2012 Feb 16. PMID 22336776
- [Result] Bondonno CP, Downey LA, Croft KD, Scholey A, Stough C, Yang X, Considine MJ, Ward NC, Puddey IB, Swinny E, Mubarak A, Hodgson JM. The acute effect of flavonoid-rich apples and nitrate-rich spinach on cognitive performance and mood in healthy men and women. Food Funct. 2014 May;5(5):849-58. doi: 10.1039/c3fo60590f. PMID 24676365
- [Result] Callahan BJ, McMurdie PJ, Rosen MJ, Han AW, Johnson AJ, Holmes SP. DADA2: High-resolution sample inference from Illumina amplicon data. Nat Methods. 2016 Jul;13(7):581-3. doi: 10.1038/nmeth.3869. Epub 2016 May 23. PMID 27214047
- [Result] Cole JR, Wang Q, Fish JA, Chai B, McGarrell DM, Sun Y, Brown CT, Porras-Alfaro A, Kuske CR, Tiedje JM. Ribosomal Database Project: data and tools for high throughput rRNA analysis. Nucleic Acids Res. 2014 Jan;42(Database issue):D633-42. doi: 10.1093/nar/gkt1244. Epub 2013 Nov 27. PMID 24288368
- [Result] Parks DH, Chuvochina M, Waite DW, Rinke C, Skarshewski A, Chaumeil PA, Hugenholtz P. A standardized bacterial taxonomy based on genome phylogeny substantially revises the tree of life. Nat Biotechnol. 2018 Nov;36(10):996-1004. doi: 10.1038/nbt.4229. Epub 2018 Aug 27. PMID 30148503